CLINICAL TRIAL: NCT04157998
Title: Ultrasound Assessment of Metoclopramide Effect on Gastric Volume in Patients Undergoing Cesarean Section: A Randomized, Double-blind, Cross-sectional Study"
Brief Title: Ultrasound Assessment of Metoclopramide Effect on Gastric Volume in Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Collaborators: Esam Hamed (Unknown); Wafaa Hamza (Unknown)
Responsible Party: Principal Investigator, Rasha Hamed, lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 17300323
Record Dates: First submitted 2019-11-02; First posted 2019-11-08 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Aspiration Pneumonia
MeSH Terms: conditions — Pneumonia, Aspiration | interventions — Saline Solution; Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Placebo Comparator): patient receive 10 ml normal saline intravenous
  Interventions: Drug: normal saline
- metoclopramide group (Active Comparator): patient receive 10 mg metoclopramide intravenously diluted in 10 mL saline 0.9%.
  intravenous
  Interventions: Drug: Metoclopramide 10mg

INTERVENTIONS:
Drug: normal saline — intrvenous administration of 10ml normal saline preoperative
  Arms: control
Drug: Metoclopramide 10mg — intrvenous administration of 10mg metoclopramide diluted in 10ml normal saline preoperative
  Arms: metoclopramide group

SUMMARY:
the risk of aspiration pneumonitis during cesarean sections has significantly decreased. Nevertheless, precaution against gastric aspiration is still vital in patients in whom regional anesthesia contraindicated or in whom general anesthesia has to be administered (for example; during emergency cesarean delivery). The administration of intravenous anesthetics reduces the level of consciousness of a patient that compromises the protective reflexes of the upper airways. Moreover, a high level of sedation also reduces the tone of the LES (lower oesophageal sphincter). Both these situations predispose the risk of aspiration pneumonia in patients awaiting surgical interventions in supine position under general anesthesia

DETAILED DESCRIPTION:
Since regional anesthesia has largely replaced general anesthesia, the risk of aspiration pneumonitis during cesarean sections has significantly decreased. Nevertheless, precaution against gastric aspiration is still vital in patients in whom regional anesthesia contraindicated or in whom general anesthesia has to be administered (for example; during emergency cesarean delivery). The administration of intravenous anesthetics reduces the level of consciousness of a patient that compromises the protective reflexes of the upper airways. Moreover, a high level of sedation also reduces the tone of the LES (lower oesophageal sphincter). Both these situations predispose the risk of aspiration pneumonia in patients awaiting surgical interventions in supine position under general anesthesia .

The risk of aspiration increases in outpatients if the volume of the gastric contents increases beyond 25 ml, and its pH falls below 2.5. However, the risk of aspiration significantly decreases in "fasted" outpatients. Since most patients awaiting elective surgery remains fasted, routine prophylaxis for preventing aspiration pneumonitis not recommended anymore. Studies suggest that metoclopramide, in combination with H2-receptor antagonists (such as cimetidine), significantly reduces the risk of postoperative emesis and aspiration pneumonitis. However, the time available for administering oral prophylaxis with such anti-emetic and anti-histaminic is too short for these medications to be effective

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* age range between 20 to 38 years
* provided informed consent to participate.

Exclusion Criteria:

* patient refusal
* associated co-morbidity as diabetes mllitus, hypertension, preeclampsia, renal or hepatic diseases
* neurological and psychological disorders, ,
* chronic gastroesophageal reflux diseases

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant female
Enrollment: 60 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
ultrasound quantitative assessment of gastric antrum cross-sectional area | 10 hours
  gastric antrum cross-sectional area calculated as a function of the anteroposterior (APD) and craniocaudal diameter (CCD). Calculation of the cross-sectional area (CSA) conducted as a product of APD and CCD in square centimeters.
the gastric antrum cross-sectional area | 10 hours
  based on three grading system which was as follows: G-0: Antrum was flat and empty in a supine and right lateral position
  * G-1: Antrum had fluid in the right lateral position but empty in the supine position
  * G-2: Antrum had fluid and food in both the supine and right lateral position.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes